CLINICAL TRIAL: NCT05476731
Title: Phenotypic and Genotypic Characterization of Malassezia Species Isolated From Malassezia Associated Skin Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Abozaid, Demonstrator of microbiology and immunology Faculty of Medicine_ SohagUniversity, Sohag University
Other Study IDs: soh-Med-22-07-08
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Malassezia Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case
  Interventions: Diagnostic Test: culture and antifungal sensitivity and molecular detection
- control
  Interventions: Diagnostic Test: culture and antifungal sensitivity and molecular detection

INTERVENTIONS:
Diagnostic Test: culture and antifungal sensitivity and molecular detection — Samples will be cultured on Modified Dixon media for 10 days at temperature between 32-34°C.Molecular detection of malassezia species by Restriction Fragment Length Polymorphism (RFLP) .
  Antifungal susceptibility testing of the isolates will be performed using the following antifungals Fluconazole, AmphotericinB and Fluocytosine

SUMMARY:
Genus Malassezia includes 14 species, namely M. furfur, M. sympodialis, M. globosa, M. restricta, M. slooffiae, M. obtusa, M. dermatis, M. japonica and M. yamatoensis associated with normal human flora but can also cause skin lesions, and M. pachydermatis, M. nana, M. equina, M. caprae and M. cuniculiare associated with animals. Few studies found that M. pachydermatis may be transmitted to humans from pets. M. pachydermmatis is the only lipid independent species while others are lipid dependent .

As Malassezia species have similar morphological and biochemical features, the currently used phenotypic techniques for diagnosis of Pityriasis versicolor usually do not allow rapid and exact characterization. In addition; they are time-consuming, multi-step processes requiring several experimental methods. Therefore, several molecular typing methods have been used successfully, resulting in identification and classification of new Malassezia species

Aim of the work:

1. Phenotypic and Genotypic Characterization of Malassezia Species.
2. Identify antifungal resistance pattern among isolated fungus.

ELIGIBILITY:
Inclusion Criteria:

Characteristic lesions of hypopigmented or hyperpigmented scaly macules and patches which may be associated with itching in patients with Pityriasis versicolor and scales of Seborrheic dermatitis and scales from patients with Atopic dermatitis.

Exclusion Criteria:

Patients with skin lesions of extensive desquamation or inflammation that do not match Pityriasis versicolor , Seborrheic dermatitis or Atopic dermatitis. Patients who had received topical antifungal therapy within last three months or oral antifungal therapy within the last six months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Characteristic lesions of hypopigmented or hyperpigmented scaly macules and patches which may be associated with itching in patients with Pityriasis versicolor and scales of Seborrheic dermatitis and scales from patients with Atopic dermatitis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
frequency of malassezia in patients | 6 months
  frequency of malassezia in patients with malassezia associated skin infection

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Angiolella L, Carradori S, Maccallini C, Giusiano G, Supuran CT. Targeting Malassezia species for Novel Synthetic and Natural Antidandruff Agents. Curr Med Chem. 2017;24(22):2392-2412. doi: 10.2174/0929867324666170404110631. PMID 28393697
- [Background] Gaitanis G, Magiatis P, Hantschke M, Bassukas ID, Velegraki A. The Malassezia genus in skin and systemic diseases. Clin Microbiol Rev. 2012 Jan;25(1):106-41. doi: 10.1128/CMR.00021-11. PMID 22232373
- [Background] Lee YW, Byun HJ, Kim BJ, Kim DH, Lim YY, Lee JW, Kim MN, Kim D, Chun YJ, Mun SK, Kim CW, Kim SE, Hwang JS. Distribution of malassezia species on the scalp in korean seborrheic dermatitis patients. Ann Dermatol. 2011 May;23(2):156-61. doi: 10.5021/ad.2011.23.2.156. Epub 2011 May 27. PMID 21747613
- [Background] Lyakhovitsky A, Shemer A, Amichai B. Molecular analysis of Malassezia species isolated from Israeli patients with pityriasis versicolor. Int J Dermatol. 2013 Feb;52(2):231-3. doi: 10.1111/j.1365-4632.2012.05595.x. PMID 23347312